CLINICAL TRIAL: NCT05504057
Title: Evaluation of Treatments With Antihistamines and Amantadine in the Evolution of the SARS-CoV-2 Infection
Brief Title: Antihistamines, Amantadine and Evolution of the SARS-CoV-2 Infection
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Principal Investigator, Anna Puigdellívol-Sánchez, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: 02-22-161-060
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: antihistamines; amantadine; hospital admissions; survival
MeSH Terms: conditions — COVID-19 | interventions — Histamine Antagonists; Amantadine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with chronic treatment with antihistamines or amantadine: The % of patients having antihistamines or amantadine as chronic treatment that suffered COVID would be compared to the population of the Terrassa Health Consortium (THC) of the same age groups.
  Interventions: Drug: Antihistamine; Drug: Amantadine
- Other population of the THC: The % of patients of the Terrassa Health Consortium that suffered COVID19 infection of the same age groups.

INTERVENTIONS:
Drug: Antihistamine — Observation of the rate of COVID19 infection, the rate of hospitalization, the rate of survival and postcovid syndrome and thrombosis among patients previously treated with antihistamines
  Other Names: Antihistamine as crhonic treatment and COVID19 infection.
  Groups: Patients with chronic treatment with antihistamines or amantadine
Drug: Amantadine — Observation of the rate of COVID19 infection, the rate of hospitalization, the rate of survival and the rate of postcovid syndrome and thrombosis among patients previously treated with amantadine
  Other Names: Amantadine as chronic treatment and COVID19 infection.
  Groups: Patients with chronic treatment with antihistamines or amantadine

SUMMARY:
The rates of symptomatic COVID19 infection, hospital admission among COVID19 cases and survival would be quantified in patiens chronically treated with antihistamines or amantadine, with the aim of determining the role of antihistamines and amantadine in the evolution of COVID19.

DETAILED DESCRIPTION:
BACKGROUND: According to previous reports, all 84 eldery residents in nuersing homes in Yespes (Toledo, Spain), had a 100% of positive serology for COVID-19 in June 2020, but none died nor hospitalized after receiving early treatment with antihistamines. Other case reports have suggested a protective role of amantadine, since infected patients showed a very mild COVID19 infection.

OBJECTIVES.Determine the role of antihistamines and amantadine in the evolution of COVID19.

METHODS. Describe the rate of hospitalization, ICU, survival, postcovid syndrome and thrombosis among COVID 19 cases having antihistamines and amantadine as chronic treatments.

The rates would be stratified by age groups and compared with the same age groups of the population assigned to the public free Access Terrassa Health Consortium.

ELIGIBILITY:
Inclusion Criteria: Patients having chronic treatment with antihistamines or amantadine -

Exclusion Criteria: None

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population assigned to the Public and free Access Terrassa Health Consortium
Sampling Method: Non-Probability Sample
Enrollment: 140660 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
Hospital Admissions. | from march 2020.
  Rate of Hospitalization among COVID 19 infections

SECONDARY OUTCOMES:
Survival | from march 2020
  Survival among COVID1 hospitalized cases.
Symptomatic infection | from march 2020
  Patients suffering a symptomatic COVID19 infection within a determinate age group
Postcovid syndrome | from april 2020
  Patients developing postcovid syndrome after COVID19 infection
Thrombosis | from april 2020
  Patients developing thrombosis (with particular assessment of stroke, cardiac infarction, retinal vessels and pulmonary embolism)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Puigdellívol, PhD, Principal Investigator — Terrassa Health Consortium
Locations (2):
- Spain (2):
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital of Terrassa, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
Once the papers related to the study are published, a statement will be included offering data when contacting with the authors.

REFERENCES:
- [Background] Moran Blanco JI, Alvarenga Bonilla JA, Homma S, Suzuki K, Fremont-Smith P, Villar Gomez de Las Heras K. Antihistamines and azithromycin as a treatment for COVID-19 on primary health care - A retrospective observational study in elderly patients. Pulm Pharmacol Ther. 2021 Apr;67:101989. doi: 10.1016/j.pupt.2021.101989. Epub 2021 Jan 16. PMID 33465426
- [Background] Cortes-Borra A, Aranda-Abreu GE. Amantadine in the prevention of clinical symptoms caused by SARS-CoV-2. Pharmacol Rep. 2021 Jun;73(3):962-965. doi: 10.1007/s43440-021-00231-5. Epub 2021 Feb 18. PMID 33604795
- [Result] Puigdellivol-Sanchez A, Juanes-Gonzalez M, Calderon-Valdiviezo A, Losa-Puig H, Valls-Foix R, Gonzalez-Salvador M, Lozano-Paz C, Vidal-Alaball J. COVID-19 in Relation to Chronic Antihistamine Prescription. Microorganisms. 2024 Dec 13;12(12):2589. doi: 10.3390/microorganisms12122589. PMID 39770791
- [Result] Puigdellivol-Sanchez A, Juanes-Gonzalez M, Calderon-Valdiviezo A, Valls-Foix R, Gonzalez-Salvador M, Lozano-Paz C, Vidal-Alaball J. COVID-19 in Relation to Polypharmacy and Immunization (2020-2024). Viruses. 2024 Sep 27;16(10):1533. doi: 10.3390/v16101533. PMID 39459868